CLINICAL TRIAL: NCT03387293
Title: Effect of Food Insulin Index on Metabolic Parameters in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Zeynep Caferoglu, PhD, Assistant Professor Doctor, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 116S069
Record Dates: First submitted 2017-12-12; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Pediatric Obesity
Keywords: Pediatric Obesity; Insulin Resistance; Diet
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LGI-LII Breakfast (Experimental): Low glycemic index, low insulin index (LGI-LII) breakfast as a test meal
  Interventions: Other: LGI-LII Breakfast; Other: LGI-HII Breakfast
- LGI-HII Breakfast (Experimental): Low glycemic index, high insulin index (LGI-HII) breakfast as a test meal
  Interventions: Other: LGI-LII Breakfast; Other: LGI-HII Breakfast

INTERVENTIONS:
Other: LGI-LII Breakfast — This test meal with low GI and low FII amounts were served as a breakfast after 12-hours fasting and participants were asked to consume the meal in full, within 15 min.
Other: LGI-HII Breakfast — In crossover design, this test meal with low GI and high FII amounts were served as a breakfast to compare the LGI-LII Breakfast.

SUMMARY:
The aim of this study was to determine the effect of food insulin index (FII) on metabolic parameters and appetite in obese adolescents with insulin resistance. A randomized, single-blind and crossover trial included 15 obese adolescents aged 12-18 years with insulin resistance. All participants were submitted two different breakfasts: low glycemic index, low insulin index (LGI-LII) and low glycemic index, high insulin index (LGI-HII), with a 1-week washout period between meals. At time 0 (just before breakfast), 15, 30, 45, 60, 90, 120, 180 and 240 minutes after the meal, serum glucose, insulin and c-peptide levels were measured and appetite was evaluated by visual analog scale. At the end of four hours, participants were served ad libitum lunch meal. Then, the foods eaten at lunch were recorded and their energy and nutrient analysis was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-18 years
* Age- and sex-specific body mass index (BMI) ≥95th percentile of the World Health Organization (WHO) growth-reference data
* New diagnosis and not receiving any treatment
* Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) >3.16

Exclusion Criteria:

* Hypertension, cardiovascular disease, diabetes mellitus or any other significant metabolic, endocrine or gastrointestinal disease
* Use of tobacco or alcohol
* Taking any medications
* Having difficulties for physical activity

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose response | Four hours postprandial period (from fasting to 240 minutes after the test breakfast)
  Postprandial glucose response was quantified as area under the curve (AUC) (mg/dL x minutes), which was calculated according to the trapezoidal rule by using serum glucose values at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes.
Postprandial insulin response | Four hours postprandial period
  Postprandial insulin response was quantified as AUC (μU/mL x minutes), which was calculated according to the trapezoidal rule by using serum insulin values at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes.
Postprandial C-peptide response | Four hours postprandial period
  Postprandial C-peptide response was quantified as AUC (ng/mL x minutes), which was calculated according to the trapezoidal rule by using serum C-peptide values at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes.

SECONDARY OUTCOMES:
Hunger rating | Four hours postprandial period
  Visual analogue scale (VAS) ratings were measured by using a question "How hungry do you feel? (not at all hungry - as hungry as I ever felt)" at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes, and hunger rating was quantified as AUC (mm x minutes), which was calculated according to the trapezoidal rule by using those VAS scores.
Fullness rating | Four hours postprandial period
  Visual analogue scale (VAS) ratings were measured by using a question "How full do you feel? (not at all full - totally full)" at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes, and fullness rating was quantified as AUC (mm x minutes), which was calculated according to the trapezoidal rule by using those VAS scores.
Desiring to eat | Four hours postprandial period
  Visual analogue scale (VAS) ratings were measured by using a question "How strong is your desire to eat? (very weak - very strong)" at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes, and desiring to eat was quantified as AUC (mm x minutes), which was calculated according to the trapezoidal rule by using those VAS scores.
Prospective food consumption | Four hours postprandial period
  Visual analogue scale (VAS) ratings were measured by using a question "How much do you think you can eat? (no food at all - a large amount of food)" at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes, and prospective food consumption was quantified as AUC (mm x minutes), which was calculated according to the trapezoidal rule by using those VAS scores.
Desiring for sweet | Four hours postprandial period
  Visual analogue scale (VAS) ratings were measured by using a question "Would you like to eat something sweet? (No, not at all - Yes, very much)" at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes, and desiring for sweet was quantified as AUC (mm x minutes), which was calculated according to the trapezoidal rule by using those VAS scores.
Desiring for salty | Four hours postprandial period
  Visual analogue scale (VAS) ratings were measured by using a question "Would you like to eat something salty? (No, not at all - Yes, very much)" at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes, and desiring for salty was quantified as AUC (mm x minutes), which was calculated according to the trapezoidal rule by using those VAS scores.
Desiring for savoury | Four hours postprandial period
  Visual analogue scale (VAS) ratings were measured by using a question "Would you like to eat something savoury? (No, not at all - Yes, very much)" at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes, and desiring for savoury was quantified as AUC (mm x minutes), which was calculated according to the trapezoidal rule by using those VAS scores.
Desiring for fatty | Four hours postprandial period
  Visual analogue scale (VAS) ratings were measured by using a question "Would you like to eat something fatty? (No, not at all - Yes, very much)" at time points 0, 15, 30, 45, 60, 90, 120, 180 and 240 minutes, and desiring for fatty was quantified as AUC (mm x minutes), which was calculated according to the trapezoidal rule by using those VAS scores.
Subsequent energy consumption | Four hours after consuming test meal (at 240 minutes)
  At 240 minutes after the test breakfast, participants were presented with an ad libitum lunch following appetite sensation measurement. Participants selected from a buffet-style meal. During the lunch, participants were left alone in a quiet room with controlled lightning and ambient room temperature, and asked to consume whatever they wanted and to eat until they felt comfortably full. Foods were weighted or measured to the nearest 0.1 g before consumption, and any remaining food was reweighed to determine intake at lunch. Energy intake was calculated using The National Food Composition Database (TurKomp) and manufacturer labelling.
Visual appeal of test meal | Immediately after consuming test meal (at 15 minutes)
  Visual analogue scale (VAS) ratings were measured by using a question "How is the visual appeal of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal).
Smell of test meal | Immediately after consuming test meal (at 15 minutes)
  Visual analogue scale (VAS) ratings were measured by using a question "How is the smell of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal).
Taste of test meal | Immediately after consuming test meal (at 15 minutes)
  Visual analogue scale (VAS) ratings were measured by using a question "How is the taste of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal).
Aftertaste of test meal | Immediately after consuming test meal (at 15 minutes)
  Visual analogue scale (VAS) ratings were measured by using a question "Is there any perceived taste in your mouth after test meal? (Much - None)" at time points 15 minutes (immediately after consuming test meal).
Palatability of test meal | Immediately after consuming test meal (at 15 minutes)
  Visual analogue scale (VAS) ratings were measured by using a question "How is the palatability of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal).

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT03387293/Prot_SAP_000.pdf